CLINICAL TRIAL: NCT03275155
Title: The PAthophysiology and Risk of Atrial Fibrillation Detected After Ischemic StrokE (PARADISE): Prospective Non-interventional Cohort Study
Brief Title: Pathophysiology and Risk of Atrial Fibrillation Detected After Ischemic Stroke
Acronym: PARADISE
Status: Active, not recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Western University, Canada (Other); London Health Sciences Centre (Other); Parkwood Hospital, London, Ontario (Other); El Instituto de Neurociencia Cognitiva y Traslacional (INCYT) (Unknown); Instituto de Neurologia Cognitiva (INECO) (Unknown)
Responsible Party: Sponsor
Other Study IDs: R-17-032
Record Dates: First submitted 2017-08-24; First posted 2017-09-07 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Stroke, Ischemic; Transient Ischemic Attack; Atrial Fibrillation
Keywords: Autonomic Dysfunction; Inflammation; Cognitive impairment; Interoception; Gait impairment
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient; Atrial Fibrillation; Primary Dysautonomias; Inflammation; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- AFDAS: patients without history of atrial fibrillation before the qualifying stroke or transient ischemic attack who are diagnosed with atrial fibrillation during the 14 days of monitoring
- KAF: atrial fibrillation known before the stroke or transient ischemic attack
- NSR: patients without a history of atrial fibrillation who do not develop atrial fibrillation during the 14 days of cardiac monitoring

SUMMARY:
This prospective non-interventional cohort study investigates the pathophysiology of Atrial Fibrillation Detected After Stroke or transient ischemic attack (AFDAS) by comparing the autonomic function and inflammation between patients with AFDAS, patients with atrial fibrillation (AF) diagnosed before the ischemic event or known AF (KAF), and patients with normal sinus rhythm (NSR) after 14 day of cardiac monitoring following the event onset.

DETAILED DESCRIPTION:
This study enrolls patients with acute ischemic stroke at the London Health Sciences Center in London, Ontario, Canada. The heart rhythm of the patients is monitored with a CardioSTAT® Holter device (Icentia) for 14 days after the ischemic event onset. Based on this cardiac monitoring and previous medical history, patients are stratified into three groups: (a) atrial fibrillation detected after stroke or transient ischemic attack (AFDAS), (b) atrial fibrillation diagnosed before the ischemic event or known AF (KAF), and (c) normal sinus rhythm (NSR).

Autonomic function is assessed by the levels of plasma catecholamines, a battery of validated autonomic tests [autonomic reflex screening (ARS)], heart rate variability (HRV) through data obtained by Holter monitoring by standard quantitative analysis methods according to the guidelines of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology and by the analysis of diurnal variation of heart rate. Blood samples are collected for the analysis of inflammatory markers (e.g. CRP, TNF-α, IL-1β, and IL-6), and potential AFDAS predictors such as brain natriuretic peptide (BNP- AFDAS biomarker), endothelin-1 (endothelial dysfunction marker), Lipoprotein(a) [Lp(a)] and thrombin-activatable fibrinolysis inhibitor (TAFI) plasma levels, TAFI activity, TAFI single nucleotide polymorphisms (SNPs), apo(a) isoform size and plasma catecholamines levels. Furthermore, specific neuroimaging findings (e.g., specific regions of the insula or its connections) and clinical features (e.g., impaired interoceptive processing, cognitive impairment, etc) are also analyzed. Interoception is assessed using a heartbeat detection task without feedback condition and gait, balance, frailty, and cognitive status in patients are evaluated by the administration of a battery of tests. Stroke recurrence will be assessed by a structured phone interview at 6 and 12 months after the initial stroke.

ELIGIBILITY:
Inclusion Criteria:

1. MCA territory-transient ischemic attack or -acute ischemic stroke patients seen in the Emergency Department or admitted to University Hospital, London, Ontario, Canada
2. Age ≥ 18 years old
3. Patient or Substitute Decision Maker must give written informed consent

Exclusion Criteria:

1. Patients with autonomic dysfunction such as Parkinson's disease that can be interfering with outcome assessment based on qualified investigator's judgment.
2. Patients taking tricyclic antidepressant (TCAs)
3. Patients in whom the acute stroke is primarily hemorrhagic
4. Patients with both TIA and atrial fibrillation
5. Patients with both TIA and large vessel disease
6. Patients with inflammatory diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ischemic stroke and transient ischemic attack patients presenting at the University Hospital of the London Health Science Center, London, Ontario, Canada.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-04-18 (Actual); Primary Completion 2026-05-07 (Estimated); Study Completion 2026-05-07 (Estimated)

PRIMARY OUTCOMES:
Changes and Differences in Autonomic Function | Within 48 hours of stroke onset and at 12, 30 and 90 days.
  Differences in Composite Autonomic Severity Score (CASS) on an 11-point scale between patients with (a) AFDAS, (b) KAF , and (c) NSR
Changes and Differences in Inflammatory Responses | Within 48 hours of stroke onset and at 12, 30 and 90 days.
  Differences in levels of plasma markers or temporal responses (CRP,TNFα, IL-6, IL-1β, etc) between patients with (a) AFDAS, (b)KAF and (c) NSR.
Changes and Differences in Heart Rate Variability (HRV) | At 14 days.
  Differences in HRV parameters between patients with (a) AFDAS, and (b) NSR

SECONDARY OUTCOMES:
Biomarkers | Within 48 hours of stroke onset, at 12, 30 and 90 days and at 6 months.
  Differences in levels of plasma markers (BNP,endothelin-1, Lp(a), and TAFI) or neuroimaging/clinical predictors between patients with (a) AFDAS , (b) KAF and (c) NSR
Atrial Fibrillation Burden | At 14 days
  Difference in atrial fibrillation burden (sum of atrial fibrillation episodes for a period of time) of AFDAS subjects with mild stroke/TIA compared to AFDAS subjects with moderate/severe stroke.
Gait Impairments | At 6 months
  Differences in gait parameters in patients with a) AFDAS , (b) KAF and (c) NSR.
Frailty | At 6 months
  Differences in frailty in patients with (a) AFDAS , (b) KAF and (c) NSR
Cognitive Impairment | At 6 months
  Differences in cognition in patients with (a) AFDAS , (b) KAF and (c) NSR

OTHER OUTCOMES:
Stroke Recurrence | At 90, 180, and 360 days
  Number of stroke recurrences in patients with (a) AFDAS , (b) KAF and (c) NSR
Death | At 90, 180, and 360 days
  Number of deaths in (a) AFDAS , (b) KAF and (c) NSR groups

CONTACTS AND LOCATIONS:
Overall Officials: Luciano A Sposato, MD, Principal Investigator — Lawson Health Research Institute, London Health Sciences Center, Western University
Locations (1):
- University Hospital, London Helath Sciences Center, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No